CLINICAL TRIAL: NCT00756704
Title: The Effectiveness of Smoking Cessation Guidelines in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R21DA021607 (NIH); R21DA021607 (NIH)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Cigarette Smoking
Keywords: Smoking Cessation; Emergency Medicine; Emergency Nursing; Effectiveness Trial; Implementation; Relapse prevention
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baseline Period (No Intervention)
- Intervention Period (Experimental)
  Interventions: Behavioral: Smoking cessation guideline implementation

INTERVENTIONS:
Behavioral: Smoking cessation guideline implementation — 1. a tutorial on brief cessation counseling for ED nurses and physicians
  2. use of an ED algorithm that includes recommended tobacco counseling items
  3. fax referral of motivated smokers to Quitline Iowa for proactive telephone counseling plus free nicotine replacement therapy
  4. group feedback to ED staff
  Arms: Intervention Period

SUMMARY:
Although 78% of smokers report that a health professional has previously advised them to quit smoking, most smokers are not advised to stop smoking or offered assistance with smoking cessation during a given ED visit. There are multiple barriers to routine implementation of smoking cessation guidelines by emergency clinicians, however, and rigorously performed clinical trials are needed to demonstrate that routine screening and counseling of ED patients results in increased quit rates. To determine the feasibility of implementing the Agency for Healthcare Research and Quality (AHRQ) Smoking Cessation Guideline in the ED, we will conduct a clinical trial in 974 ambulatory adult smokers who present to 2 emergency departments, using a pre-post design. During the 3-month baseline period, clinicians will perform their usual duties but will not receive training in use of the AHRQ Guideline. Based on the Chronic Care Model, the 3-month intervention period will include: 1) a tutorial on brief cessation counseling for ED nurses and physicians, 2) use of an ED algorithm that includes recommended tobacco counseling items, 3) fax referral of motivated smokers to Quitline Iowa for proactive telephone counseling plus free nicotine replacement therapy, and 4) group and individual feedback to ED staff. We will conduct exit interviews of ED patients to assess performance of guideline-recommended actions by ED staff and 3- and 6-month telephone follow-up to determine 7-day point-prevalence abstinence (with biochemical confirmation of self-reported quitters at 6 months). Our main analyses will examine the contrast between the intervention and control periods in the performance of guideline-recommended actions and in 6-month quit rates, using hierarchical logistic regression to adjust for baseline differences in potentially confounding patient variables. In secondary analyses, we will assess the change in attitudes of ED nurses and physicians toward smoking cessation counseling. This feasibility study will determine the receptivity of patients and ED staff to the guideline-based intervention and will provide estimates of effect size in planning a full scale multi-site clinical trial of the study intervention in community hospital EDs.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the Emergency Department by private vehicle or on a walk-in basis
* Current cigarette smoker (5 or more cigarettes per day)

Exclusion Criteria:

* Acute medical decompensation (e.g., acute respiratory failure requiring intubation, cardiac arrest, cardiogenic or septic shock)
* Life-threatening trauma
* Altered mental status
* Dementia
* Language barrier
* Incarceration
* Transfer to another ED
* Departure from the ED prior to evaluation
* Inability to be contacted by telephone
* ED presentation for sexual assault
* ED presentation for acute psychiatric crisis (e.g., suicidal ideation)
* Participation in a smoking cessation program in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Performance of smoking cessation guideline-recommended actions by ED staff | Assessed within two weeks after discharge from ED

SECONDARY OUTCOMES:
7-day point-prevalence smoking abstinence | 3 and 6 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: David A Katz, MD, MSc, Principal Investigator — The Univesity of Iowa College of Medicine
Locations (2):
- United States (2):
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - The University of Iowa Hospitals and Clinics Emergency Treatment Center, Iowa City, Iowa

REFERENCES:
- [Result] Katz D, Vander Weg M, Nugent A, Kim R, Graham M, Holman J, Hillis S, Titler M. Adherence to smoking cessation guidelines in the emergency department. J Gen Intern Med 2009; 24 (Suppl 1): S15.
- [Derived] Katz DA, Paez MW, Reisinger HS, Gillette MT, Weg MW, Titler MG, Nugent AS, Baker LJ, Holman JE, Ono SS. Implementation of smoking cessation guidelines in the emergency department: a qualitative study of staff perceptions. Addict Sci Clin Pract. 2014 Jan 24;9(1):1. doi: 10.1186/1940-0640-9-1. PMID 24460974
- [Derived] Katz DA, Holman JE, Nugent AS, Baker LJ, Johnson SR, Hillis SL, Tinkelman DG, Titler MG, Vander Weg MW. The emergency department action in smoking cessation (EDASC) trial: impact on cessation outcomes. Nicotine Tob Res. 2013 Jun;15(6):1032-43. doi: 10.1093/ntr/nts219. Epub 2012 Nov 2. PMID 23125437